CLINICAL TRIAL: NCT03650725
Title: Evaluation of Information Provided to Patients Provided About Bowel Preparation for Morning Colonoscopy
Brief Title: Evaluation of Information on Bowel Preparation for Morning Colonoscopy
Status: Completed | Type: Observational
Sponsor: Harminder Singh (Other)
Responsible Party: Sponsor-Investigator, Harminder Singh, Associate Professor of Medicine, University of Manitoba
Organization: University of Manitoba (Other)
Other Study IDs: H2018:202
Record Dates: First submitted 2018-08-15; First posted 2018-08-29 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Colonoscopy; Patient Compliance
Keywords: Colonoscopy; bowel preparation
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mandatory Split bowel preparation: Patients will be advised to take 4 liters of polyethylene glycol (PEG), split into two 2 liter doses. The first 2 liters are to be taken starting at 1800 hours the day before the colonoscopy, and the second dose is to be taken starting 4-5 hours prior to the scheduled time for the colonoscopy. Each dose will be taken within a 2-hour time span.
  Interventions: Other: Mandatory Split bowel preparation
- Optional Split bowel preparation: Patients will be advised on split-dose bowel preparation (as per option 1), but will also receive instructions on day before bowel preparation. The instructions will indicate that split-dose bowel preparation is the optimal preparation for cleansing the bowel and for visualizing polyps, but they may choose day before bowel preparation if the split dose preparation is too difficult for them.

INTERVENTIONS:
Other: Mandatory Split bowel preparation — Intervention describes the standard of care patient split bowel preparation instructions as mandatory, instead of giving patient instructions with option of choice between split or day before bowel prep.
  Other Names: Instructions for Bowel preparation before colonoscopy
  Groups: Mandatory Split bowel preparation

SUMMARY:
Background: In randomized controlled trials, split-dose bowel preparation for colonoscopy has been shown to provide better bowel cleansing than day before bowel preparation. However, people who volunteer to be in clinical trials may be more adherent to a challenging bowel preparation regimen than people in the general community undergoing colonoscopy. This may be especially true for colonoscopies scheduled for the morning, when the later dose of the split-dose bowel preparation would be administered in the early morning hours. Hence the results of the available trials may not be applicable to patients undergoing morning colonoscopy in routine medical practices.

Aims: To compare the effectiveness of mandatory split-dose bowel preparation to optional split-dose bowel preparation protocols for morning colonoscopies in a non-inferiority pragmatic trial.

Anticipated results and significance: The study will produce a better understanding of the most effective approach to bowel preparation for early morning colonoscopies and suggest specific recommendations for colonoscopy practice.

DETAILED DESCRIPTION:
Patient will be randomized by the central booking office. Patient experience survey will be administered prior to colonoscopy. Chart review will be done to obtain data from the medical records and endoscopy reports. Please see outcomes and planned analysis.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Must have colonoscopy appointment with any 4 of the participating GI doctors at Health Sciences Centre-Winnipeg
* Must use 4 liter type of bowel preparation

Exclusion Criteria:

* Has colonoscopy appointment with non-participating GI doctor and/or a non-participating endoscopy hospital/clinic
* Patient and/or referral doctor requested a non-4 liter bowel preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Description of Population: We will enroll all persons who are scheduled to undergo colonoscopy by one of the four participating gastroenterologists at an outpatient hospital-based endoscopy centre in Winnipeg, Canada, in this trial. These four gastroenterologists have been in practice for 10 years or greater, and all perform over 400 colonoscopies annually. Patients are referred to these gastroenterologists by a centralized referral program, which is responsible for scheduling the procedure and for distributing the bowel preparation instructions- This program is randomly assigning to mandatory and optional split preparation as part of routine care; stratified randomization by early vs. later morning.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of bowel cleanliness as measured by Boston Bowel Preparation Scale Score (0-2) in all segments | At the scheduled colonoscopy procedure performed with the instructions provided, expected average within 3 months
  Proportion with adequate cleansing as measured by Boston Bowel Preparation Scale Score ≥2 in all segments. Boston Bowel Preparation Scale Score is reported as score of 0 to 3 in 3 segments of the colon. The score is then summed for a total score of 0 to 9. Higher Boston score, better quality of bowel cleanliness.

SECONDARY OUTCOMES:
Composite with any of the following: cancellations in the day before colonoscopy; no shows for colonoscopy appointment; phone calls for questions on the bowel preparation and/or rescheduling because of the bowel preparation. | Anytime before the scheduled colonoscopy procedure performed with the instructions provided, expected average within 3 months
  Determine the proportion with any of the following: cancellations in the day before colonoscopy; no shows for colonoscopy appointment (composite and separate analysis for these 2 outcomes); phone calls for questions on the bowel preparation and/or rescheduling because of the bowel preparation (indicator of staff workload generated).. This is a composite measure of number of individuals in each of the listed categories. Each will also be reported separately.
Amount of laxative intake | In the 24 hours before the scheduled colonoscopy,expected average within 3 months
  Amount of laxative intake before colonoscopy will be compared in the two groups.
Proportion with split dose laxative intake | In the 24 hours before the scheduled colonoscopy,expected average within 3 months
  Split dose refers to taking half the dose of the laxative day before colonoscopy and half on the day of the colonoscopy.
Endoscopic Outcome 1: Cecal intubation (colonoscopy completion) | At the scheduled colonoscopy procedure, expected average within 3 months
  Compare cecal intubation rate between the groups.
Endoscopic Outcome 2: Withdrawal time during colonoscopy performance | At the scheduled colonoscopy procedure, expected average within 3 months
  Compare withdrawal time between the groups.
Endoscopic Outcome 3: total time for performance of colonoscopy | At the scheduled colonoscopy procedure, expected average within 3 months
  Compare total procedure time between the groups.
Endoscopic Outcome 4: polyps during colonoscopy | At the scheduled colonoscopy procedure, expected average within 3 months
  Compare polyp detection (adenoma, sessile serrated polyps) detection rates between the groups.
Patient experience data outcome 1: use of split dose bowel preparation | Before scheduled colonoscopy procedure, expected average within 3 months
  We will determine the proportion reporting: use of split dose and day before bowel preparation
Patient experience data outcome 2: complete intake of all of the prescribed laxative | Before scheduled colonoscopy procedure, expected average within 3 months
  We will determine the proportion reporting consumption of all of the laxative
Patient experience data outcome 3: incontinence episodes while preparing for colonoscopy | Before scheduled colonoscopy procedure, expected average within 3 months
  We will determine the proportion reporting incontinence episodes during bowel preparation and during travel to the colonoscopy appointment
Patient experience data outcome 4: Sleep in night before colonoscopy | Before scheduled colonoscopy procedure, expected average within 3 months
  We will determine and compare the total duration of sleep
Patient experience data outcome 5: willingness to repeat colonoscopy using same laxative preparation | Assessed immediately before scheduled colonoscopy procedure, expected average within 3 months
  We will determine the proportion reporting patient willingness to repeat colonoscopy using same preparation
Patient experience data outcome 6: pre-colonoscopy anxiety (Likert scale 1-5) | Assessed immediately before scheduled colonoscopy procedure, expected average within 3 months
  We will determine and compare the pre-colonoscopy anxiety rating, assessed on 5 point Likert scale (1-5). Higher values represent higher anxiety.
Patient experience data outcome 7: difficulty with bowel preparation (Likert scale 1-10) | Assessed immediately before scheduled colonoscopy procedure, expected average within 3 months
  We will determine and compare difficulty with bowel preparation rating, as reported by patients on a ten point Likert scale (1-10). Higher values represent less difficulty (i.e. more tolerance)

OTHER OUTCOMES:
Quality of bowel cleanliness as measured by total Ottawa Bowel Preparation Scale Score (0-14) | At the scheduled colonoscopy procedure performed with the instructions provided, expected average within 3 months
  Ottawa Bowel Scale score is calculated as a sum of scores in the 3 segments of colon (0-4) plus amount of fluid (0-2). All of the scores in the segments will be recorded and then summed. Comparison will be as continuous variable as dichotomous score ≤ 7. Lower the score on Ottawa scale, better the cleansing quality.

CONTACTS AND LOCATIONS:
Overall Officials: Harminder Singh, MD, MPH, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Center, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rex DK. Optimal bowel preparation--a practical guide for clinicians. Nat Rev Gastroenterol Hepatol. 2014 Jul;11(7):419-25. doi: 10.1038/nrgastro.2014.35. Epub 2014 Apr 1. PMID 24686267
- [Background] Martel M, Barkun AN, Menard C, Restellini S, Kherad O, Vanasse A. Split-Dose Preparations Are Superior to Day-Before Bowel Cleansing Regimens: A Meta-analysis. Gastroenterology. 2015 Jul;149(1):79-88. doi: 10.1053/j.gastro.2015.04.004. Epub 2015 Apr 8. PMID 25863216
- [Background] Horton N, Garber A, Hasson H, Lopez R, Burke CA. Impact of Single- vs. Split-Dose Low-Volume Bowel Preparations on Bowel Movement Kinetics, Patient Inconvenience, and Polyp Detection: A Prospective Trial. Am J Gastroenterol. 2016 Sep;111(9):1330-7. doi: 10.1038/ajg.2016.273. Epub 2016 Jul 5. PMID 27377521
- [Background] Radaelli F, Paggi S, Hassan C, Senore C, Fasoli R, Anderloni A, Buffoli F, Savarese MF, Spinzi G, Rex DK, Repici A. Split-dose preparation for colonoscopy increases adenoma detection rate: a randomised controlled trial in an organised screening programme. Gut. 2017 Feb;66(2):270-277. doi: 10.1136/gutjnl-2015-310685. Epub 2015 Dec 9. PMID 26657900
- [Background] Bucci C, Rotondano G, Hassan C, Rea M, Bianco MA, Cipolletta L, Ciacci C, Marmo R. Optimal bowel cleansing for colonoscopy: split the dose! A series of meta-analyses of controlled studies. Gastrointest Endosc. 2014 Oct;80(4):566-576.e2. doi: 10.1016/j.gie.2014.05.320. Epub 2014 Jul 19. PMID 25053529
- [Background] Siddiqui AA, Yang K, Spechler SJ, Cryer B, Davila R, Cipher D, Harford WV. Duration of the interval between the completion of bowel preparation and the start of colonoscopy predicts bowel-preparation quality. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):700-6. doi: 10.1016/j.gie.2008.09.047. PMID 19251013
- [Background] Johnson DA, Barkun AN, Cohen LB, Dominitz JA, Kaltenbach T, Martel M, Robertson DJ, Boland CR, Giardello FM, Lieberman DA, Levin TR, Rex DK; US Multi-Society Task Force on Colorectal Cancer. Optimizing adequacy of bowel cleansing for colonoscopy: recommendations from the US multi-society task force on colorectal cancer. Gastroenterology. 2014 Oct;147(4):903-24. doi: 10.1053/j.gastro.2014.07.002. No abstract available. PMID 25239068
- [Background] Hassan C, Bretthauer M, Kaminski MF, Polkowski M, Rembacken B, Saunders B, Benamouzig R, Holme O, Green S, Kuiper T, Marmo R, Omar M, Petruzziello L, Spada C, Zullo A, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2013;45(2):142-50. doi: 10.1055/s-0032-1326186. Epub 2013 Jan 18. PMID 23335011
- [Background] Ton L, Lee H, Taunk P, Calderwood AH, Jacobson BC. Nationwide variability of colonoscopy preparation instructions. Dig Dis Sci. 2014 Aug;59(8):1726-32. doi: 10.1007/s10620-014-3262-8. Epub 2014 Jul 2. PMID 24985353
- [Background] Clark BT, Protiva P, Nagar A, Imaeda A, Ciarleglio MM, Deng Y, Laine L. Quantification of Adequate Bowel Preparation for Screening or Surveillance Colonoscopy in Men. Gastroenterology. 2016 Feb;150(2):396-405; quiz e14-5. doi: 10.1053/j.gastro.2015.09.041. Epub 2015 Oct 9. PMID 26439436
- [Background] Calderwood AH, Schroy PC 3rd, Lieberman DA, Logan JR, Zurfluh M, Jacobson BC. Boston Bowel Preparation Scale scores provide a standardized definition of adequate for describing bowel cleanliness. Gastrointest Endosc. 2014 Aug;80(2):269-76. doi: 10.1016/j.gie.2014.01.031. Epub 2014 Mar 12. PMID 24629422
- [Background] Parmar R, Martel M, Rostom A, Barkun AN. Validated Scales for Colon Cleansing: A Systematic Review. Am J Gastroenterol. 2016 Feb;111(2):197-204; quiz 205. doi: 10.1038/ajg.2015.417. Epub 2016 Jan 19. PMID 26782820
- [Background] Menees SB, Kim HM, Wren P, Zikmund-Fisher BJ, Elta GH, Foster S, Korsnes S, Graustein B, Schoenfeld P. Patient compliance and suboptimal bowel preparation with split-dose bowel regimen in average-risk screening colonoscopy. Gastrointest Endosc. 2014 May;79(5):811-820.e3. doi: 10.1016/j.gie.2014.01.024. Epub 2014 Mar 13. PMID 24631492
- [Background] Singh H, Kaita L, Taylor G, Nugent Z, Bernstein C. Practice and documentation of performance of colonoscopy in a central Canadian health region. Can J Gastroenterol Hepatol. 2014 Apr;28(4):185-90. doi: 10.1155/2014/635932. PMID 24729991
- [Background] Porostocky P, Chiba N, Colacino P, Sadowski D, Singh H. A survey of sedation practices for colonoscopy in Canada. Can J Gastroenterol. 2011 May;25(5):255-60. doi: 10.1155/2011/783706. PMID 21647459
- [Background] Singh H, Nugent Z, Demers AA, Kliewer EV, Mahmud SM, Bernstein CN. The reduction in colorectal cancer mortality after colonoscopy varies by site of the cancer. Gastroenterology. 2010 Oct;139(4):1128-37. doi: 10.1053/j.gastro.2010.06.052. Epub 2010 Jun 20. PMID 20600026
- [Background] Singh H, Penfold RB, De Coster C, Au W, Bernstein CN, Moffatt M. Predictors of serious complications associated with lower gastrointestinal endoscopy in a major city-wide health region. Can J Gastroenterol. 2010 Jul;24(7):425-30. doi: 10.1155/2010/714591. PMID 20652157
- [Background] Loftus R, Nugent Z, Graff LA, Schumacher F, Bernstein CN, Singh H. Patient satisfaction with the endoscopy experience and willingness to return in a central Canadian health region. Can J Gastroenterol. 2013;27(5):259-66. doi: 10.1155/2013/615206. PMID 23712300
- [Background] Singh H, Bay D, Ip S, Bernstein CN, Nugent Z, Gheorghe R, Wightman R. Pathological reassessment of hyperplastic colon polyps in a city-wide pathology practice: implications for polyp surveillance recommendations. Gastrointest Endosc. 2012 Nov;76(5):1003-8. doi: 10.1016/j.gie.2012.07.026. PMID 23078924
- [Background] Pruthi D, Duerksen DR, Singh H. The practice of gastrostomy tube placement across a Canadian regional health authority. Am J Gastroenterol. 2010 Jul;105(7):1541-50. doi: 10.1038/ajg.2009.756. Epub 2010 Jan 26. PMID 20104220
- [Background] Singh H, Turner D, Xue L, Targownik LE, Bernstein CN. Risk of developing colorectal cancer following a negative colonoscopy examination: evidence for a 10-year interval between colonoscopies. JAMA. 2006 May 24;295(20):2366-73. doi: 10.1001/jama.295.20.2366. PMID 16720822
- [Derived] Shaffer SR, Lambert P, Unruh C, Harland E, Helewa RM, Decker K, Singh H. Optimizing Timing of Follow-Up Colonoscopy: A Pilot Cluster Randomized Trial of a Knowledge Translation Tool. Am J Gastroenterol. 2024 Mar 1;119(3):547-555. doi: 10.14309/ajg.0000000000002542. Epub 2023 Oct 3. PMID 37787644
- [Derived] Dolovich C, Unruh C, Moffatt DC, Loewen C, Kaita B, Barkun AN, Martel M, Singh H. Mandatory vs. optional split-dose bowel preparation for morning colonoscopies: a pragmatic noninferiority randomized controlled trial. Endoscopy. 2023 Sep;55(9):822-835. doi: 10.1055/a-2070-5561. Epub 2023 Apr 6. PMID 37023789